CLINICAL TRIAL: NCT00659464
Title: Use of Multi-site Near Infrared Spectroscopy (NIRS) Monitoring for Hemodynamic Assessment During Tilt Table Testing in Children
Brief Title: Multi-Site Near Infrared Spectroscopy (NIRS) Monitoring of Children During Tilt Table Testing
Acronym: NIRS & Tilt
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, John Hambrook, Assistant Professor, Pediatrics Cardiology, Medical College of Wisconsin
Other Study IDs: CHW 08/22
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Syncope
Keywords: Infrared Spectroscopy; Syncope; Tilt Table Testing
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Children who present to the heart center exercise stress lab for investigation of syncope

SUMMARY:
PURPOSE OF THE STUDY

This study will explore the use of multi-site NIRS monitoring during tilt table testing, combining somatic and cerebral saturations data with hemodynamic data to establish the non-invasive assessment of global cardiac output distribution trends.

HYPOTHESIS / SPECIFIC AIMS

Study Aims: To evaluate the utility of multi-site NIRS monitoring in the cardiovascular hemodynamic assessment of children and adolescents during tilt table testing by establishing a non-invasive method to predict cardiac output maldistribution with the use of two-site NIRS monitoring in children and adolescents with syncope.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 7 and 21 years
* Referred to the exercise stress lab due to syncope

Exclusion Criteria:

* Under 7 or over 21 years of age
* Referred to the exercise stress lab for anything other than syncope

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children ages 7 through 21 years who present to exercise stress lab for investigation of syncope.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Rao, MD, Principal Investigator — Medical College of Wisconsin/Children's Hospital of Wisconsin; John Hambrook, MD, Principal Investigator — Medical College of Wisconsin/Children's Hospital of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Result] Rao RP, Danduran MJ, Dixon JE, Frommelt PC, Berger S, Zangwill SD. Near infrared spectroscopy: guided tilt table testing for syncope. Pediatr Cardiol. 2010 Jul;31(5):674-9. doi: 10.1007/s00246-010-9683-z. Epub 2010 Mar 4. PMID 20204346